CLINICAL TRIAL: NCT06080893
Title: The Effect of Preoperative Ferric Carboxymaltose Administration on Mortality in Geriatric Hip Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Özkaya, Assistant İnvestigator, Istanbul University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Istanbul Faculty of Medicine
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hip Fractures; Anemia; Complication,Postoperative
Keywords: administration, intravenous; aged; anemia / complications; anemia / drug therapy; ferric compounds; hip fractures / mortality; hip fractures / surgery
MeSH Terms: conditions — Hip Fractures; Anemia; Postoperative Complications | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric Carboxymaltose - Administrated Group (Experimental): Patients eligible for inclusion who received preop FCM intravenous therapy
  FCM will be administered intravenously at preop 24th hour according to weight and preop hgb level
  Interventions: Drug: Ferric carboxymaltose
- Ferric Carboxymaltose - Not Administrated Group (No Intervention): Patients eligible for inclusion who are not received preop FCM intravenous therapy

INTERVENTIONS:
Drug: Ferric carboxymaltose — FCM can be administered in a short IV infusion of 15-20 minutes, allowing doses of 2 g in a single session, and furthermore, FCM is excellently tolerated and safe for patients.
  FCM will be administered intravenously at preop 24th hour according to weight and preop hgb level
  Other Names: Ferinject
  Arms: Ferric Carboxymaltose - Administrated Group

SUMMARY:
Hip fractures (HF) are the most common and serious pathology affecting the hip and are associated with a high mortality risk in elderly patients. The prevalence of HF is increasing day by day and surgery is often required for its treatment. Perioperative anemia not only hinders the early recovery and rapid rehabilitation of elderly patients, but also adversely increases the need for blood transfusion, prolongs hospital length of stay (HLS) and even increases the risk of death. Although the blood transfusion threshold is restrictive, approximately one or two thirds of elderly patients with hip fracture surgery (HFS) require blood transfusion during hospitalization, and blood transfusion also has potential side effects.The most important factor in the development of anemia in HF is blood loss; however, there are other mechanisms (renal failure, inflammation, iatrogenic hemodilution) that lead to the selection of different therapeutic approaches.Oral or intravenous iron supplementation is a well-accepted alternative to counteract or prevent perioperative anemia, stimulate erythropoiesis and increase Hgb level in elderly patients. However, there are few studies addressing the relationship between iron therapy and clinical outcomes or mortality. Because ferric carboxymaltose (FCM) allows doses of 2 g in a single session (and can be administered by a short IV infusion of 15-20 minutes), and furthermore, FCM is excellently tolerated and safe for patients. This study was planned to investigate the relationship between FCM supplementation and blood transfusion volume, HLS, postoperative infection and mortality.

DETAILED DESCRIPTION:
In the prospective randomized controlled study, a 6 - 12 month follow-up of participants undergoing hip fracture surgery with and without preoperative FCM treatment will be performed. Planning is being made with a total of 200 participants from 100 participants each in the experimental and control groups. Participants over the age of 65 who are diagnosed with hip fracture at Istanbul University Istanbul Faculty of Medicine Orthopedics and Traumatology Clinic will be included in the study. Participants who meet the inclusion criteria will be randomized into 2 groups as participants with and without preopaerative FCM (20 min iv infusion) so as to evaluate laboratory values during hospital stay, perop and postop ES transfusion needs, post-discharge 6th week Hgb value and 6th and 12th month mortality information. The parameters to be examined in clinical controls in the study are age, gender, smoking, comorbidities if any, hip fracture type, surgical treatment, ASA score, body mass index, preop/postop/pre-discharge/6th week Hgb value, perop/postop transfusion amount, preop INR value and 6th month/12th month mortality status.

ELIGIBILITY:
Inclusion Criteria:

* >65 years

Exclusion Criteria:

* < 65 years
* Tumor-induced pathological fractures
* Patients undergoing preop ES replacement
* Ferric Carboxymaltose drug allergy
* Multiple trauma
* Receiving iron therapy in any form at the time of application
* Those who cannot come to postop clinical follow-up (out of town, etc.)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 209 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Mortality | 6th and 12th months
  6th and 12th month mortality information

CONTACTS AND LOCATIONS:
Overall Officials: Mert Ballı, Study Chair — Istanbul Faculty of Medicine
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Department Orthopaedics and Traumatology, Istanbul, Çapa / Fatih, Turkey (Türkiye)

REFERENCES:
- [Result] Jones JJ, Mundy LM, Blackman N, Shwarz M. Ferric Carboxymaltose for Anemic Perioperative Populations: A Systematic Literature Review of Randomized Controlled Trials. J Blood Med. 2021 May 26;12:337-359. doi: 10.2147/JBM.S295041. eCollection 2021. PMID 34079413
- [Result] Clemmensen SZ, Kragholm KH, Melgaard D, Hansen LT, Riis J, Cavallius C, Morch MM, Krogager ML. Association between intravenous iron therapy and short-term mortality risk in older patients undergoing hip fracture surgery: an observational study. J Orthop Surg Res. 2021 May 18;16(1):320. doi: 10.1186/s13018-021-02462-x. PMID 34006287
- [Result] Parker MJ. Iron supplementation for anemia after hip fracture surgery: a randomized trial of 300 patients. J Bone Joint Surg Am. 2010 Feb;92(2):265-9. doi: 10.2106/JBJS.I.00883. PMID 20124051
- [Result] Bernabeu-Wittel M, Romero M, Ollero-Baturone M, Aparicio R, Murcia-Zaragoza J, Rincon-Gomez M, Monte-Secades R, Melero-Bascones M, Rosso CM, Ruiz-Cantero A; PAHFRAC-01 Investigators. Ferric carboxymaltose with or without erythropoietin in anemic patients with hip fracture: a randomized clinical trial. Transfusion. 2016 Sep;56(9):2199-211. doi: 10.1111/trf.13624. Epub 2016 May 14. PMID 27195774
- [Result] Bernabeu-Wittel M, Aparicio R, Romero M, Murcia-Zaragoza J, Monte-Secades R, Rosso C, Montero A, Ruiz-Cantero A, Melero-Bascones M; PAHFRAC-01 investigators. Ferric carboxymaltose with or without erythropoietin for the prevention of red-cell transfusions in the perioperative period of osteoporotic hip fractures: a randomized contolled trial. The PAHFRAC-01 project. BMC Musculoskelet Disord. 2012 Feb 21;13:27. doi: 10.1186/1471-2474-13-27. PMID 22353604
- [Result] Munoz M, Gomez-Ramirez S, Auerbach M. Stimulating erythropoiesis before hip fracture repair for reducing blood transfusion: should we change the hemoglobin cutoff level for defining anemia in females? Transfusion. 2016 Sep;56(9):2160-3. doi: 10.1111/trf.13750. No abstract available. PMID 27624208